CLINICAL TRIAL: NCT04423588
Title: Prospective, Monocentric Study of Dexlansoprazole Absorption Preoperative and 6 and 12 Months After Proximal Roux-en-Y Gastric Bypass Surgery and of the Incidence of Marginal Ulcers 6 and 12 Months After Surgery
Brief Title: Dexlansoprazole Absorption and Marginal Ulceration After Gastric Bypass
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: Spital Limmattal Schlieren (Other)
Responsible Party: Principal Investigator, Prof Urs Zingg, Prof. Dr. med. Urs Zingg, Spital Limmattal Schlieren
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-02326
Record Dates: First submitted 2020-02-07; First posted 2020-06-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Bariatric Surgery
Keywords: Proton Pump Inhibitor
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dexlansoprazole (Other): The PPI Dexilant (active substance: dexlansoprazole) is administered to the study participants in a prophylactic Regimen for 6 months after the PRYGB-surgery. This drug is already approved by Swissmedic and on the markets in Switzerland. The dosage is 1 capsule 60 mg per os daily in the morning.
  Interventions: Diagnostic Test: dexlansoprazole serum concentration; Diagnostic Test: upper endoscopy

INTERVENTIONS:
Diagnostic Test: dexlansoprazole serum concentration — 6 blood samples are collected at fixed time Points after oral Administration of 1 dose of dexilant at regular patients visits preoperatively and 3 and 6 months post-surgery.
Diagnostic Test: upper endoscopy — 6 and 12 months after surgery the occurrence of marginal ulcers in the same Patient Group is examined by upper endoscopy. The 12-month endoscopy is part of the Routine postoperative diagnosis, the 6-month endoscopy is for study purpose.

SUMMARY:
In Switzerland, the most commonly performed bariatric procedure is the proximal Roux-en-y gastric Bypass surgery. Since marginal ulceration is a known complication after this Operation, a Proton pump Inhibitor (PPI) prophylaxis is prescribed postoperatively. Bariatric surgery may have an impact on the absorption and consequently on the efficacy of drugs. There are only very little data on the pharmacokinetics of PPIs following PRYGB.

The aim of this study is to analyze the serum concentration of dexlansoprazole preoperative and after PRYGB surgery in patients taking PPI prophylaxis and to examine the incidence of marginal ulcers postoperatively in the same population.

DETAILED DESCRIPTION:
This prospective, monocentric study includes 30 patients undergoing a proximal Roux-en-Y gastric Bypass surgery and receiving 6 months of postoperative PPI prophylaxis with Dexilant (dexlansoprazole). The aim is to examine if the LPRYGB has an impact on the absorption of dexlansoprazole. Peripheral blood samples from the study participants are obtained at fixed time points after oral Administration of a capsule Dexilant preoperatively as well as 3 and 6 months after surgery. The incidence of marginal ulceration in the same patient population is assessed by upper endoscopy 6 and 12 months after surgery. The surgery, the PPI prophylaxis and the upper endoscopy 12 months post-surgery aren't for study purpose. Data collection is made by measuring serum drug concentration, patient questionnaires, pill count and upper endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for study and surgery as documented by signature
* Male and Female Patients over 18 years old eligible for bariatric surgery at the Department of General Surgery, Limmattal Hospital, according to criteria of the Swiss Study Group for Morbid Obesity (SMOB) and international Guidelines
* BMI ≥ 35
* Failure of conservative Treatment for 2 years
* Type of surgery: LPRYGB
* Helicobacter pylori negative
* Smoker (≥ 1 cigarette daily)
* Women in reproductive Age: negative pregnancy test

Exclusion Criteria:

* Contraindication for a bariatric surgery according to SMOB-criteria
* Contraindication for PPIs
* Pregnant or breastfeeding women
* Pre- or intraoperative decision for other type of surgery than LPRYGB
* Active malignancy
* Chronic liver disease Child-Pugh B or C
* Abuse of drugs or alcohol
* Suspect of non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change of dexlansoprazole Serum concentration | 3 months
  Determination of the dexlansoprazole concentration (ng/ml) in the participants blood at time 0, 60, 90, 120, 210, 300 min after having swallowed a Dosis of dexilant preoperatively and 3 months after surgery
Change of dexlansoprazole Serum concentration | 6 months
  Determination of the dexlansoprazole concentration (ng/ml) in the participants blood at time 0, 60, 90, 120, 210, 300 min after having swallowed a Dosis of dexilant preoperatively and 6 months after surgery

SECONDARY OUTCOMES:
Incidence of Marginal ulceration | 6 months
  Study of the incidence of marginal ulcers in the participants 6 months after surgery
Incidence of Marginal ulceration | 12 months
  Study of the incidence of marginal ulcers in the participants 12 months after surgery
Incidence of Marginal ulceration | 6 months
  Study of the incidence of marginal ulcers in participants undergoing a upper endoscopy in the presence of symptoms Prior to the end of the 6 post-operative months

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, Prof. Dr. med., Principal Investigator — Chefarzt Chirurgie, Limmattal Hospital